CLINICAL TRIAL: NCT01867216
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Ascending Oral Doses of LY2922470 in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of Multiple Doses of LY2922470 in Participants With Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14797; I6K-FW-GLEB (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-05-28; First posted 2013-06-03 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LY2922470

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Multiple oral dose of placebo administered to participants with diabetes once or twice daily for 28 days
  Interventions: Drug: Placebo
- LY2922470 (Experimental): Multiple ascending dose of LY292470 (starting at 60 mg) administered orally to participants with diabetes once or twice daily for 28 days
  Interventions: Drug: LY2922470

INTERVENTIONS:
Drug: Placebo — Administered orally as capsules
  Arms: Placebo
Drug: LY2922470 — Administered orally as capsules
  Arms: LY2922470

SUMMARY:
The main purpose of this study is to determine the safety of LY2922470, taken as oral capsules, once or twice daily for approximately 28 days, in participants with diabetes. It also aims to determine how long the drug stays in the body and how it affects blood sugar levels. A screening appointment is required within 28 days before the start of the study and a follow up appointment is required approximately 14 days after the last study dose is taken.

ELIGIBILITY:
Inclusion Criteria:

* Must be a male, or a female who cannot become pregnant, and who has type 2 diabetes
* Have a glycated hemoglobin (HbA1c) value of greater than or equal to 6.5% and less than or equal to 11% at screening
* Do not have any change to their diabetes treatment (exercise with or without metformin) for at least 4 weeks prior to screening
* Have a screening body mass index (BMI) of 18.0 to 45.0 kilograms per square meter (kg/m^2)
* Have blood pressure, pulse rate, blood and urine laboratory test results acceptable for the study

Exclusion Criteria:

* Are currently participating in another clinical study or completed one in the last 30 days
* Have a history of significant heart, lung, liver, kidney, stomach or brain disease, or have any medical problems which may cause an increased risk during the study
* Have electrocardiogram (ECG) readings that are not suitable for the study
* Are infected with hepatitis B or hepatitis C
* Are infected with human immunodeficiency virus (HIV)
* Have donated blood equal to or more than 500 mL within 56 days before the first dose of drug or have donated plasma within 7 days before the first dose or provided any blood donation within the last month from screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chula Vista, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eatontown, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo QD or BID: Placebo administered orally once daily (QD) or twice daily (BID) for up to 28 days.
- 60 mg LY2922470 QD: 60 mg LY2922470 administered orally QD for up to 28 days.
- 200 mg LY2922470 QD: 200 mg LY2922470 administered orally QD for up to 28 days.
- 500 mg LY2922470 QD: 500 mg LY2922470 administered orally QD for up to 28 days.
- 1200 mg LY2922470 QD: 1200 mg LY2922470 administered orally QD for up to 28 days.
- 150 mg LY2922470 BID: 150 mg LY2922470 administered orally BID for up to 28 days.
- 400 mg LY2922470 BID: 400 mg LY2922470 administered orally BID for up to 28 days.
Period: Overall Study
Arm/Group | Placebo QD or BID | 60 mg LY2922470 QD | 200 mg LY2922470 QD | 500 mg LY2922470 QD | 1200 mg LY2922470 QD | 150 mg LY2922470 BID | 400 mg LY2922470 BID
Started | 16 | 8 | 8 | 8 | 9 | 8 | 9
Received Study Drug | 14 | 8 | 8 | 8 | 9 | 8 | 9
Completed | 12 | 8 | 8 | 8 | 8 | 8 | 8
Not Completed | 4 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unable to Place Catheter for Blood Draws | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Placebo QD or BID: Placebo administered orally QD or BID for up to 28 days.
- Total: Total of all reporting groups
Arm/Group | Placebo QD or BID | 60 mg LY2922470 QD | 200 mg LY2922470 QD | 500 mg LY2922470 QD | 1200 mg LY2922470 QD | 150 mg LY2922470 BID | 400 mg LY2922470 BID | Total
Number analyzed (Participants) | 14 | 8 | 8 | 8 | 9 | 8 | 9 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (9.9) | 59.9 (6.6) | 52.8 (8.0) | 58.6 (7.8) | 59.8 (7.6) | 54.0 (6.4) | 50.2 (9.3) | 54.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 1 | 4 | 4 | 4 | 22
  Male | 10 | 6 | 5 | 7 | 5 | 4 | 5 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 1 | 1 | 2 | 4 | 5 | 6 | 27
  Not Hispanic or Latino | 6 | 7 | 7 | 6 | 5 | 3 | 3 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 3 | 5 | 5 | 5 | 3 | 3 | 1 | 25
  White | 11 | 3 | 3 | 3 | 6 | 5 | 7 | 38
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 8 | 8 | 8 | 9 | 8 | 9 | 64
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m²)] — BMI is an estimate of body fat based on body weight divided by height squared.
  kilograms per square meter (kg/m²) | 31.00 (4.86) | 28.10 (3.19) | 30.76 (3.74) | 31.08 (3.40) | 30.20 (6.56) | 34.36 (4.04) | 32.90 (6.08) | 31.19 (4.89)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] — HbA1c is a form of hemoglobin that is primarily measured to identify the average plasma glucose concentration over prolonged periods of time.
  percentage of glycosylated hemoglobin | 8.29 (1.08) | 8.58 (1.48) | 7.74 (1.29) | 7.91 (1.69) | 7.24 (0.49) | 8.09 (1.25) | 7.96 (1.21) | 7.99 (1.24)
Fasting Blood Glucose [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 145.92 (50.50) | 128.45 (39.38) | 132.39 (37.09) | 140.19 (49.53) | 137.11 (26.19) | 149.50 (38.40) | 149.56 (44.21) | 141.05 (40.99)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline through Study Completion (up to 56 days)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD or BID | 60 mg LY2922470 QD | 200 mg LY2922470 QD | 500 mg LY2922470 QD | 1200 mg LY2922470 QD | 150 mg LY2922470 BID | 400 mg LY2922470 BID
Number analyzed (Participants) | 14 | 8 | 8 | 8 | 9 | 8 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC) From Time Zero to 24 Hours Postdose (AUC[0-24]) of LY2922470
Time Frame: Day 1: Predose, 0.5, 1.5, 2.5, 4, 6, 12, 16, 24 hours postdose and Day 28: Predose, 0.5, 1.5, 2.5, 4, 6, 12, 16, 24 hours postdose
Population: All participants who received LY2922470 and had sufficient evaluable AUC(0-24) values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | 60 mg LY2922470 QD | 200 mg LY2922470 QD | 500 mg LY2922470 QD | 1200 mg LY2922470 QD | 150 mg LY2922470 BID | 400 mg LY2922470 BID
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 9
nanograms*hour/milliliter (ng*h/mL)
  Day 1 | 4220 (52) | 11,600 (27) | 25,100 (30) | 81,400 (34) | 21,000 (47) | 50,700 (45)
  Day 28: number analyzed (Participants) | 8 | 7 | 5 | 8 | 8 | 8
  Day 28 | 5660 (31) | 15,300 (43) | 25,000 (47) | 65,300 (49) | 21,300 (51) | 44,800 (38)

3. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY2922470
Time Frame: Day 1: Predose, 0.5, 1.5, 2.5, 4, 6, 12, 16, 24 hours postdose and Day 28: Predose, 0.5, 1.5, 2.5, 4, 6, 12, 16, 24, 48 hours postdose
Population: All participants who received LY2922470 and had sufficient evaluable Cmax values. For BID arms, Cmax from time 0-6 hours.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 60 mg LY2922470 QD | 200 mg LY2922470 QD | 500 mg LY2922470 QD | 1200 mg LY2922470 QD | 150 mg LY2922470 BID | 400 mg LY2922470 BID
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 9
ng/mL
  Day 1 | 723 (39) | 1540 (23) | 2750 (42) | 8200 (38) | 1510 (54) | 3150 (58)
  Day 28: number analyzed (Participants) | 8 | 7 | 5 | 8 | 8 | 8
  Day 28 | 1070 (32) | 1630 (70) | 3410 (33) | 7900 (49) | 1540 (42) | 2980 (37)

4. Secondary Outcome: Pharmacokinetics: Time to Maximum Concentration (Tmax) of LY2922470
Time Frame: as for outcome 3
Population: All participants who received LY2922470 and had sufficient evaluable Tmax values. For BID arms, Tmax from time 0-6 hours.
Measure: Median (Full Range); unit: hours
Arm/Group | 60 mg LY2922470 QD | 200 mg LY2922470 QD | 500 mg LY2922470 QD | 1200 mg LY2922470 QD | 150 mg LY2922470 BID | 400 mg LY2922470 BID
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 9
hours
  Day 1 | 1.50 [1.50 to 2.50] | 2.50 [1.50 to 4.00] | 2.75 [1.50 to 16.0] | 4.00 [1.50 to 6.00] | 2.00 [1.50 to 4.00] | 2.50 [1.50 to 4.00]
  Day 28: number analyzed (Participants) | 8 | 7 | 5 | 8 | 8 | 9
  Day 28 | 1.50 [1.50 to 1.50] | 3.92 [1.50 to 6.00] | 1.50 [1.50 to 2.50] | 2.50 [1.50 to 6.00] | 1.51 [1.50 to 4.00] | 1.50 [1.50 to 4.00]

5. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Day 28
Time Frame: Baseline, Day 28
Population: All participants who received study drug and had sufficient evaluable HbA1c values.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Placebo QD or BID | 60 mg LY2922470 QD | 200 mg LY2922470 QD | 500 mg LY2922470 QD | 1200 mg LY2922470 QD | 150 mg LY2922470 BID | 400 mg LY2922470 BID
Number analyzed (Participants) | 12 | 8 | 8 | 8 | 8 | 8 | 8
percentage of glycosylated hemoglobin | -0.38 (0.45) | -0.54 (0.32) | -0.43 (0.58) | -0.24 (0.52) | -0.16 (0.67) | -0.34 (0.38) | 0.01 (0.44)

6. Secondary Outcome: Change From Baseline in Blood Glucose Area Under the Effective Concentration Curve (AUEC₀-₂₄) During Mixed Meal Tolerance Test at Day 28
Time Frame: Day 28: Predose, 0.5,1.5, 2.5, 4, 6, 12, 16, 24 hours Postdose
Population: All participants who received study drug and had sufficient evaluable blood glucose values.
Measure: Mean (Standard Deviation); unit: mg*h/dL
Arm/Group | Placebo QD or BID | 60 mg LY2922470 QD | 200 mg LY2922470 QD | 500 mg LY2922470 QD | 1200 mg LY2922470 QD | 150 mg LY2922470 BID | 400 mg LY2922470 BID
Number analyzed (Participants) | 10 | 5 | 8 | 8 | 8 | 8 | 8
mg*h/dL | 21.7 (724) | -93 (165) | 70.4 (1160) | -499 (493) | -205 (583) | -531 (549) | -621 (943)

7. Secondary Outcome: Change From Baseline in C-Peptide Area Under the Effective Concentration Curve (AUEC₀-₁₂) During Mixed Meal Tolerance Test at Day 28
Time Frame: Day 28: Predose, 0.5,1.5, 2.5, 4, 6, 12 hours Postdose
Population: All participants who received study drug and had sufficient evaluable c-peptide values.
Measure: Mean (Standard Deviation); unit: picomoles*h per liter (pmol*h/L)
Arm/Group | Placebo QD or BID | 60 mg LY2922470 QD | 200 mg LY2922470 QD | 500 mg LY2922470 QD | 1200 mg LY2922470 QD | 150 mg LY2922470 BID | 400 mg LY2922470 BID
Number analyzed (Participants) | 12 | 8 | 6 | 8 | 7 | 6 | 8
picomoles*h per liter (pmol*h/L) | 665 (4970) | 147 (3560) | 793 (4220) | -159 (3780) | -740 (2890) | 1230 (1660) | -2230 (2810)

ADVERSE EVENTS:
Description: All participants who received at least one dose of study drug.
Arm/Group | Placebo QD or BID | 60 mg LY2922470 QD | 200 mg LY2922470 QD | 500 mg LY2922470 QD | 1200 mg LY2922470 QD | 150 mg LY2922470 BID | 400 mg LY2922470 BID
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/8 | 0/8 | 0/8 | 0/9 | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 5/14 | 3/8 | 4/8 | 4/8 | 5/9 | 1/8 | 6/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo QD or BID (N=14) | 60 mg LY2922470 QD (N=8) | 200 mg LY2922470 QD (N=8) | 500 mg LY2922470 QD (N=8) | 1200 mg LY2922470 QD (N=9) | 150 mg LY2922470 BID (N=8) | 400 mg LY2922470 BID (N=9)
Asthenopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (3) | 5 (5) | 0 (0) | 3 (4)
Faeces pale (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infrequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 1 (2) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nipple disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days